CLINICAL TRIAL: NCT05639296
Title: Expert Learning in Musculoskeletal Ultrasound - the Effect of Discovery Learning
Brief Title: Expert Learning in Musculoskeletal Ultrasound
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Maya Dreier Carstensen, MD, PhD fellow, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: 2023-004
Record Dates: First submitted 2022-11-22; First posted 2022-12-06 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Musculoskeletal Diseases
Keywords: Medical education; Ultrasound
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSUS experts: Physicians with extensive experience with MSUS (performed more than 1000 examinations).
  Interventions: Other: Discovery learning (DL)

INTERVENTIONS:
Other: Discovery learning (DL) — DL makes the trainee practice before giving them instruction, "Do-Then-Tell", thereby promoting their ability to use and build upon their existing knowledge.

SUMMARY:
Musculoskeletal ultrasound (MSUS) is a complex procedure and requires lifelong theoretical and practical training to ensure continued professional development.

Currently, the teaching approach for experts in MSUS is theoretical preparation first and then hands-on training, the "Tell-Then-Do" approach. The existing literature on optimizing training for experts is sparse, and it is unknown if the training intervention Discovery Learning could be a more effective teaching method for this group of learners.

ELIGIBILITY:
Inclusion Criteria:

* Experts in MSUS, defined as physicians who have performed more than 1000 MSUS examinations

Exclusion Criteria:

* Physicians who have not performed 1000 MSUS examinations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians with a Rheumatology background. All experts in the field of MSUS.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
How do experts in MSUS approach a new and unfamiliar MSUS task? | January 2023
  All performances will be analyzed to examine how the experts solve the MSUS case, e.g., do they use the available material etc? More specifically, how much time (in seconds) do they use on different problem-solving methods such as "information seeking", "trial and error", and "systematic evaluation".

SECONDARY OUTCOMES:
How do the experts respond to DL? | January 2023
  i.e., are they comfortable changing the learning situation from "Tell-Then-Do" to "Do-Then-Tell"? The participants will fill out a post-course questionnaire. 10 questions to be answered on a 5 point Likert scale from (range 1-5).

CONTACTS AND LOCATIONS:
Overall Officials: Stine Maya Dreier Carstensen, MD, Principal Investigator — COPECARE (Copenhagen Center for Arthritis Research) Rigshospitalet, Glostrup
Locations (1):
- Barcelona University, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brydges R, Fiume A, Grierson L. Mastery versus invention learning: impacts on future learning of simulated procedural skills. Adv Health Sci Educ Theory Pract. 2022 May;27(2):441-456. doi: 10.1007/s10459-022-10094-x. Epub 2022 Mar 23. PMID 35320441
- [Background] Steenhof N, Woods NN, Van Gerven PWM, Mylopoulos M. Productive failure as an instructional approach to promote future learning. Adv Health Sci Educ Theory Pract. 2019 Oct;24(4):739-749. doi: 10.1007/s10459-019-09895-4. Epub 2019 May 14. PMID 31089856
- [Background] Terslev L, Hammer HB, Torp-Pedersen S, Szkudlarek M, Iagnocco A, D'Agostino MA, Schmidt WA, Uson J, Bruyn GA, Filippucci E, Moller I, Balint P, Wakefield R, Naredo E. EFSUMB minimum training requirements for rheumatologists performing musculoskeletal ultrasound. Ultraschall Med. 2013 Oct;34(5):475-7. doi: 10.1055/s-0033-1335143. Epub 2013 May 21. PMID 23696065